CLINICAL TRIAL: NCT06225414
Title: Empowering Hispanic Patients' Lung Cancer Screening Uptake (Empower Latinx)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Radiological Society of North America (Other)
Responsible Party: Principal Investigator, Gelareh Sadigh, Associate Professor In Residence, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 4471; UCI 23-219 (Other: CFCCC)
Record Dates: First submitted 2024-01-15; First posted 2024-01-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Screening; Multi-level intervention
MeSH Terms: conditions — Lung Neoplasms | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Enhanced Usual Care (Experimental): Usual Care + Brief Educational Material
  Interventions: Other: Usual Care; Behavioral: Brief Patient Education
- Arm B: Empower Latinx (Experimental): * PCP notifications of patients' LCS eligibility (addressing provider time constraints and barrier in identifying eligible patients);
  * Patients' education (addressing knowledge barriers);
  * Patients' referral to financial navigation resources (addressing health-related social risks)
  * Patients' reminder to discuss LCS during PCP visit.
  Interventions: Other: Usual Care; Behavioral: Patient education; Behavioral: Referral to financial navigation resources; Behavioral: Patient Reminders; Behavioral: Provider Reminders

INTERVENTIONS:
Other: Usual Care — The usual care includes a provider flag in electronic medical record (EMR) on patients' eligibility for LCS if their smoking history is complete.
Behavioral: Brief Patient Education — Brief one-page education material on lung cancer screening benefits and risk
  Arms: Arm A: Enhanced Usual Care
Behavioral: Patient education — Patients will be sent information (in preferred language) on lung cancer risk, lung cancer screening (LCS) benefits, harms, false positive rates, recommendations of follow-up for positive results, and exam insurance coverage.
  Arms: Arm B: Empower Latinx
Behavioral: Referral to financial navigation resources — Patients who self-report needing help with health-related social risks at baseline will be sent a brochure (in preferred language) from patient advocate foundation (PAF), a national non-profit financial navigation organization, where patients can self-refer.
  Arms: Arm B: Empower Latinx
Behavioral: Patient Reminders — within 2 weeks prior to appointment, patients will receive a text message or a phone call (if not having a phone that receives text messaging) encouraging patients to discuss lung cancer screening with their provider.
  Arms: Arm B: Empower Latinx
Behavioral: Provider Reminders — Within 2 weeks prior to primary care appointment, providers will be notified of their patient's eligibility for lung cancer screening and their reported barriers.
  Arms: Arm B: Empower Latinx

SUMMARY:
The Hispanic/Latinx community (hereafter Hispanic) is the country's second-largest racial/ethnic group, accounting for 19.1% of the total population. However, they remain one of the most underserved populations with suboptimal access to healthcare and screening services due to low income, lack of health insurance, perceived discrimination, language barriers, and limited health literacy. Lung cancer is the leading cause of cancer related mortality with 1.8 million annual deaths worldwide, with Hispanic patients known to have lower survival rates compared with non-Hispanic whites. Lung cancer screening (LCS) with low dose computed tomography (LDCT) decreases this mortality rate of lung cancer by 20%. Yet many Latinx patients who are eligible for lung cancer screening are still falling through the cracks which prevents patients the ability to detect lung cancer early. This study will test and compare the effect of a multi-level intervention on ordering LDCT within 4 months after patient enrollment to those in an Enhanced Usual Care. Our proposed intervention includes:

* Primary care provider notifications of patients' LCS eligibility;
* Patients' education;
* Patients' referral to financial navigation resources;
* Patients' reminder to discuss LCS during primary care provider (PCP) visit.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50- 80 years of age.
* Be able to speak English and Spanish
* Must have a Primary Care Provider.
* History of 20-pack year smoking history ( based on survey self-report)
* Current smoker or a former smoker who has quit smoking within the last 15 years (based on survey self-report)
* Resident of California

Exclusion Criteria:

* Prior history of lung cancer
* Chest CT for any reason in the last 12 months based on self-report and UCI EMR
* History of Alzheimer's disease or dementia

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2025-12-11 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with order of Low-dose CT (LDCT) for lung cancer screening (LCS) | Within 4 months of randomization

SECONDARY OUTCOMES:
Number of Participants who received LDCT for LCS | Within 4 months of randomization
Number of Participants with the documented discussion of lung cancer screening with their providers in the electronic medical record | Within 4 months of randomization
Patients' perceived risk of lung cancer | Baseline and 4 months after randomization
  3-item perceived risk of lung cancer questionnaire developed by Carter Harris et al (Cancer Nurs, 2018) will be used. The responses for each item will be based on a 5-point likert scale. A sum score will be calculated based on responses to all 3 item. Score will range between 3 and 15. Higher score= higher perceived risk.
Patients' perceived severity of lung cancer | Baseline and 4 months after randomization
  5-items about the health consequences and severity of lung cancer will be used. The responses for each item will be based on a 5-point likert scale. A sum score will be calculated based on responses to all items. Score will range between 5-25. Higher score= higher perceived benefits.
Patients' perceived benefits of lung cancer screening | Baseline and 4 months after randomization
  6-item perceived benefit of lung cancer questionnaire developed by Carter Harris et al (Cancer Nurs, 2018) will be used. The responses for each item will be based on a 5-point likert scale. A sum score will be calculated based on responses to all items. Score will range between 6-30. Higher score= higher perceived benefits.
Patients' perceived barriers of lung cancer screening | Baseline and 4 months after randomization
  19-item perceived barriers of lung cancer questionnaire will be used. 17 of these items were developed by Carter Harris et al (Cancer Nurs, 2018). The responses for each item will be based on a 5-point likert scale. A sum score will be calculated based on responses to all 17 validated items. Score will range between 17 and 85. Higher score= higher perceived barriers. An additional score including all 19 items will also be calculated.
Patients' self-efficacy of lung cancer screening | Baseline and 4 months after randomization
  10-item self-efficacy for lung cancer screening questionnaire will be used. 9 of these items were developed by Carter Harris et al (Cancer Nurs, 2018). The responses for each item will be based on a 5-point likert scale. A sum score will be calculated based on responses to all 9 validated item. Score will range between 9 and 45. Higher score= higher self-efficacy. An additional score including all 10 items will also be calculated.
Patients' knowledge about lung cancer screening | Baseline and 4 months after randomization
  9 questions adopted and modified from Volk R et al (PMID: 24518006) will be used. Responses will be based on true, false, unsure. Sum of correctly responded questions will be calculated. Higher score= higher knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Gelareh Sadigh, MD, Principal Investigator — University of California, Irvine
Locations (10):
- United States (10):
  - UCI Health Family Health Center - Anaheim, Anaheim, California
  - UCI Health-Costa Mesa, Costa Mesa, California
  - UCI Health-Irvine, Irvine, California
  - UCI Health-Laguna hilla, Laguna Hills, California
  - UCI Health-Newport, Newport Beach, California
  - UCI Health SeniorHealth Center -Pavillion 4, Orange, California
  - UCI Medical Center, Pavilion 3, Orange, California
  - UCI Health Family Health Center - Santa Ana, Santa Ana, California
  - UCI-Health Tustin, Tustin, California
  - UCI Health-Yorba Linda, Yorba Linda, California

IPD SHARING:
Plan to Share IPD: No